CLINICAL TRIAL: NCT05714202
Title: A Phase 3, Open-Label, Multi-Center, Randomized Study Evaluating the Efficacy and Safety of TAR-200 in Combination With Cetrelimab or TAR-200 Alone Versus Intravesical Bacillus Calmette-Guérin (BCG) in Participants With BCG-naïve High-Risk Non-Muscle Invasive Bladder Cancer
Brief Title: A Study of TAR-200 in Combination With Cetrelimab or TAR-200 Alone Versus Intravesical Bacillus Calmette-Guérin (BCG) in Participants With BCG-naïve High-risk Non-muscle Invasive Bladder Cancer (HR-NMIBC)
Acronym: SunRISe-3
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR109223; 17000139BLC3002 (Other: Janssen Research & Development, LLC); 2020-004506-64 (EudraCT Number); 2023-507187-39-00 (Registry Identifier: EUCT number)
Expanded Access: NCT06877676 (Approved for marketing)
Record Dates: First submitted 2023-01-27; First posted 2023-02-06 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment Group A: TAR-200 + Cetrelimab (Experimental): Participants will receive intravesical TAR-200 once every 3 weeks (Q3W) and cetrelimab.
  Interventions: Drug: TAR-200; Biological: Cetrelimab
- Treatment Group B: Bacillus Calmette-Guerin (BCG) Vesiculture (Active Comparator): Participants will receive intravesical BCG once every week for 6 weeks (induction) and then followed by once every week for 3 weeks starting at Weeks 12, 24, 48, 72, and 96 (maintenance).
  Interventions: Biological: BCG Vesiculture
- Treatment Group C: TAR-200 Alone (Experimental): Participants will receive intravesical TAR-200 alone once Q3W.
  Interventions: Drug: TAR-200

INTERVENTIONS:
Drug: TAR-200 — TAR-200 will be administered intravesically.
  Other Names: JNJ-17000139
  Arms: Treatment Group A: TAR-200 + Cetrelimab; Treatment Group C: TAR-200 Alone
Biological: Cetrelimab — Cetrelimab will be administered.
  Other Names: JNJ-63723283
  Arms: Treatment Group A: TAR-200 + Cetrelimab
Biological: BCG Vesiculture — BCG will be administered intravesically.
  Arms: Treatment Group B: Bacillus Calmette-Guerin (BCG) Vesiculture

SUMMARY:
The purpose of this study is to compare event-free survival (EFS) in participants with Bacillus Calmette-Guerin (BCG)-naive high-risk non-muscle invasive bladder cancer (HR-NMIBC), including high-grade papillary Ta, any T1, or carcinoma in situ (CIS), between TAR-200 plus cetrelimab (Group A) and TAR-200 alone (Group C) versus intravesical BCG (Group B).

DETAILED DESCRIPTION:
Bladder cancer is the tenth most common malignancy worldwide. About 75 percent (%) of bladder cancers are non-muscle invasive at diagnosis with approximately 25% of NMIBC patients have HR, NMIBC. The TAR-200/gemcitabine (JNJ-17000139) product is an intravesical drug delivery system regulated as an investigational drug. The drug constituent consists of gemcitabine and osmotic minitablets. Cetrelimab (JNJ-63723283) is a fully human immunoglobulin G4 (IgG4) kappa monoclonal antibody (mAb) that binds programmed-cell death protein (PD)-1. The mainstay of treatment for HR-NMIBC is transurethral resection of bladder tumor, followed by intravesical treatment with BCG. In this study metronomic dosing of intravesical gemcitabine, delivered via TAR-200, alone or in combination with cetrelimab will be evaluated and compared against intravesical BCG. The study consists of a Screening phase, Treatment phase, and Follow-up phase. The total duration of the study will be up to 5 years and 2 months. Efficacy, Safety, pharmacokinetics (PK), and biomarkers will be assessed at specific time points during the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed initial diagnosis by local pathology (within 90 days of the most recent signed informed consent) of high grade non-muscle invasive bladder cancer (HR-NMIBC) (high-grade Ta, any T1 or carcinoma in-situ [CIS]), in participants who are Bacillus Calmette Guérin (BCG)-naïve
* BCG-naïve (participants who have not received prior intravesical BCG or who previously received but stopped BCG more than 3 years before date of randomization are eligible)
* All visible papillary disease must be fully resected (absent) prior to date of randomization and documented at baseline cystoscopy. Local urine cytology at screening must be negative or atypical (for high-grade urothelial carcinoma [HGUC]) for patients with papillary only disease (without CIS)
* Eastern Cooperative Oncology Group (ECOG) performance status Grade 0, 1, or 2
* All adverse events associated with any prior surgery and/or intravesical therapy must have resolved to common terminology criteria for adverse events (CTCAE) version 5.0 Grade less than (<) 2 prior to date of randomization
* Participants must be willing to undergo all study procedures

Exclusion Criteria:

* Presence or history of histologically confirmed, muscle invasive, locally advanced, nonresectable, or metastatic urothelial carcinoma (that is, greater than and equal to [>=] T2)
* Must not have had urothelial carcinoma or histological variant at any site outside of the urinary bladder (that is, urethra, ureter, or renal pelvis). Ta/any T1/CIS of the upper urinary tract (including renal pelvis and ureter) is allowable if treated with complete nephroureterectomy more than 24 months prior to randomization
* Presence of any bladder or urethral anatomic feature (example, urethral stricture) that, in the opinion of the investigator, may prevent the safe insertion, indwelling use, removal of TAR-200 or administration of intravesical BCG. Participants with tumors involving the prostatic urethra in men will be excluded
* A history of clinically significant polyuria with recorded 24-hour urine volumes greater than 4000 milliliters (mL)
* Indwelling catheters are not permitted; however, intermittent catheterization is acceptable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1135 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2029-09-18 (Estimated); Study Completion 2029-09-18 (Estimated)

PRIMARY OUTCOMES:
Event-free Survival (EFS) | Up to 5 years 2 months
  EFS is defined as the time from randomization to either the time of the first recurrence of high-risk disease, progression, or death due to any cause, whichever occurs first. For participants with carcinoma In-situ (CIS), persistent disease at 6 months (Week 24) is also considered an EFS event. Progression is defined as: an increase of stage from Ta to T1 or from CIS to T1 or progression to muscle invasive bladder cancer (MIBC) (T greater than or equal to [>=] 2) or to lymph node (N+) or to distant disease (M+), whichever occurs first.

SECONDARY OUTCOMES:
Overall Complete Response (CR) Rate | Up to 5 years 2 months
  Overall CR will be measured by determining the percentage of participants with CIS who have no presence of high-risk disease at 6 months.
Duration of CR | Up to 5 years 2 months
  Duration of CR is defined from the time of first CR achieved to first evidence of recurrence, progression or death due to any cause (whichever occurs first) for participants who achieve a CR.
Recurrence-Free Survival (RFS) | Up to 5 years 2 months
  RFS is defined as the time from randomization to the time of the first recurrence of high-risk disease, or death due to any cause, whichever occurs first.
Time to Progression (TTP) | Up to 5 years 2 months
  TTP is defined as the time from randomization to the date of first documented evidence of disease progression or death due to disease progression, whichever occurs first.
Overall Survival (OS) | Up to 5 years 2 months
  OS is defined as the time from randomization to death, due to any cause.
Cancer Specific Survival (CSS) | Up to 5 years 2 months
  CSS is defined as the time from randomization to the date of death due to bladder cancer.
Number of Participants with Adverse Events (AEs) by Grades According to Common Terminology Criteria for Adverse Events (CTCAE) | Up to 5 years 2 months
  Number of participants with AEs by severity grade as assessed by CTCAE version 5 will be reported. Grade refers to the severity of AE as follows: Grade 1- Mild; Grade 2- Moderate; Grade 3- Severe; Grade 4- Life-threatening; Grade 5- Death related to adverse event.
Number of Participants with Adverse Events (AEs) | Up to 5 years 2 months
  Number of participants with AEs will be reported. An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non-investigational) product, whether or not related to that medicinal (investigational or non-investigational) product.
Number of Participants with Change from Baseline in Laboratory Abnormalities | Up to 5 years 2 months
  Number of participants with change from baseline in laboratory abnormalities will be reported. Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1- Mild, Grade 2- Moderate, Grade 3- Severe, Grade 4- Life-threatening, and Grade 5- Death related to adverse event.
Number of Participants with Change from Baseline in Vital Signs Abnormalities | Up to 5 years 2 months
  Number of participants with change from baseline in vital signs (blood pressure [systolic and diastolic], heart rate, temperature, and weight) abnormalities will be reported.
Change from Baseline in European Organisation for Research and Treatment of Cancer Quality of life Questionnaire - Non-muscle Invasive Bladder Cancer EORTC QLQ- NMIBC 24 | Up to 5 years 2 months
  EORTC QLQ-NMIBC 24 is a 24-item questionnaire for evaluating the Health-related quality of life (HRQoL) of participants with superficial (non-muscle-invasive) bladder cancer. The questionnaire is designed to supplement the quality of life questionnaire (QLQ-C30) and incorporates 6 multi-item scales and 5 single items. Ratings for each item range from 1 (not at all) to 4 (very much).
Time to Symptom Deterioration as Assessed by EORTC-QLQ-NMIBC 24 Scores | Up to 5 years 2 months
  EORTC QLQ-NMIBC 24 is a 24-item questionnaire for evaluating the HRQoL of participants with superficial (non-muscle-invasive) bladder cancer. The questionnaire is designed to supplement the QLQ-C30 and incorporates 6 multi-item scales and 5 single items. Ratings for each item range from 1 (not at all) to 4 (very much).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (240):
- United States (51):
  - Mayo Clinic, Scottsdale, Arizona
  - Arkansas Urology, Little Rock, Arkansas
  - VA Long Beach Health Care System, Long Beach, California
  - Genesis Research, LLC - West Coast Urology, Los Alamitos, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - Genesis Research, San Diego, California
  - Providence Saint Johns Cancer Institute, Santa Monica, California
  - Providence Medical Foundation, Santa Rosa, California
  - Colorado Clinical Research, Lakewood, Colorado
  - Urological Research Network, Hialeah, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - The Emory Clinic Department of Urology, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Duly Health and Care, Lisle, Illinois
  - Blessing Hospital, Quincy, Illinois
  - Urology of Indiana, Carmel, Indiana
  - First Urology, Jeffersonville, Indiana
  - AMR Kansas City Oncology, Merriam, Kansas
  - Wichita Urology Group, Wichita, Kansas
  - Chesapeake Urology Research Associates, Hanover, Maryland
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University Of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - The Urology Center, PC, Omaha, Nebraska
  - Cooper Health System MD Anderson Cancer Center at Cooper, Camden, New Jersey
  - VA NY Harbor Healthcare System, New York, New York
  - Icahn School of Medicine at Mt. Sinai, New York, New York
  - Associated Medical Professionals of Ny, Syracuse, New York
  - SUNY Upstate Med Univ, Syracuse, New York
  - Vidant Urology - Greenville, Greenville, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Central Ohio Urology Group, Gahanna, Ohio
  - Centers for Advanced Urology LLC d b a MidLantic Urology, Bala-Cynwyd, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - UPMC Shadyside Hospital, Pittsburgh, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology Associates, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Urology Austin, Austin, Texas
  - Urology Clinics of North Texas, Dallas, Texas
  - Houston Metro Urology, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Urology San Antonio Research, San Antonio, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - George E. Wahlen VAMC, Salt Lake City, Utah
  - Urology Of Virginia, Pllc, Virginia Beach, Virginia
  - Spokane Urology, Spokane, Washington
- Argentina (7):
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Sociedade Beneficente de Senhoras Hospital Sirio Libanes, Buenos Aires
  - Cemaic Centro Privado de Especialidades Medicas Ambulatorias e Investigacion Clinica, Córdoba
  - Centro Urologico Profesor Bengio, Córdoba
  - Hospital Privado Centro Medico de Cordoba, Córdoba
  - Hospital Privado de la Comunidad, Mar del Plata
  - Instituto Medico Rio Cuarto, Río Cuarto
- Australia (4):
  - Austin Health, Heidelberg
  - Macquarie University Hospital, Macquarie University
  - Hollywood Private Hospital, Nedlands
  - Mater Hospital Brisbane, South Brisbane
- Belgium (9):
  - ZNA Middelheim, Antwerp
  - AZ Sint-Jan, Bruges
  - AZ Sint-Lucas, Bruges
  - AZ Maria Middelares, Ghent
  - UZ Gent, Ghent
  - Centre Hospitalier de l'Ardenne, Libramont-Chevigny
  - AZ Delta, Roeselare
  - Vitaz, Sint-Niklaas
  - GZA Ziekenhuizen- Campus St Augustinus, Wilrijk
- Brazil (14):
  - Fundacao Pio XII, Barretos
  - NAIC Nair Antunes Instituto do Cancer, Bauru
  - Universidade Estadual De Campinas, Campinas
  - Liga Paranaense de Combate ao Cancer, Curitiba
  - Liga Norte Riograndense Contra O Cancer, Natal
  - Irmandade Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Hospital Regional do Cancer - Hospital de Esperança, Presidente Prudente
  - Hospital Sao Rafael, Salvador
  - Hospital Ana Nery Santa Cruz do Sul, Santa Cruz do Sul
  - CEPHO Centro de Estudos e Pesquisa de Hematologia e Oncologia, Santo André
  - Fundacao Faculdade de Medicina - Instituto do Cancer do Estado de Sao Paulo, São Paulo
  - Fundacao Antonio Prudente A C Camargo Cancer Center, São Paulo
  - Sociedade Beneficente Israelita Brasileira Hospital Albert Einstein, São Paulo
  - Real e Benemerita Associacao Portuguesa de Beneficencia, São Paulo
- Canada (6):
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - St Josephs Healthcare Hamilton, Hamilton, Ontario
  - Princess Margaret Cancer Centre University Health Network, Toronto, Ontario
  - CHUM - Centre hospitalier universitaire de Montreal, Montreal, Quebec
  - CHU de Quebec Universite Laval Hopital de l Enfant Jesus, Québec, Quebec
  - Unite de Recherche Clinique du CISSS des Laurentides, Saint Jerome Quebec, Quebec
- China (22):
  - Peking University First Hospital, Beijing
  - Beijing Hospital, Beijing
  - Beijing Luhe Hospital, Capital Medical University, Beijing
  - The First Bethune Hospital of Jilin University, Changchun
  - Hunan Province Cancer Hospital, Changsha
  - West China Hospital Sichuan University, Chengdu
  - Chongqing University Cancer Hospital, Chongqing
  - People's Hospital of Deyang City, Deyang
  - Sun Yat Sen University Cancer Center, Guangzhou
  - Zhejiang Provincial People's Hospital, Hangzhou
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou
  - Nanjing Drum Tower Hospital, Nanjing
  - The First Affiliated Hospital of Ningbo University, Ningbo
  - Ruijing Hospital Affiliated To Shanghai Jiaotong University School Of Medicine, Shanghai
  - Huadong Hospital Affiliated to Fudan University, Shanghai
  - Shengjing Hospital Of China Medical University, Shenyang
  - The Second Hospital Of Tianjin Medical University, Tianjin
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - TongJi Hospital of TongJi Medical College of Huazhong University of Science & Technology, Wuhan
  - First Affiliated Hospital of Medical College of Xi'an Jiaotong University, Xi'an
  - Yantai Yuhuangding Hospital, Yantai
  - Henan Cancer Hospital, Zhengzhou
- Czechia (7):
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Krajská nemocnice Liberec a.s., Liberec
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Thomayerova nemocnice, Onkologicka klinika, Prague
  - Fakultni nemocnice v Motole, Prague
- France (16):
  - Polyclinique Bordeaux Nord Acquitaine, Bordeaux
  - CHU Gabriel-Montpied, Clermont-Ferrand
  - CHU Grenoble, Grenoble
  - Polyclinique de Limoges - Francois Chenieux, Limoges
  - Hôpital Edouard Herriot, Lyon
  - CHU de Nantes hotel Dieu, Nantes
  - CHU Nimes, Nîmes
  - Centre Hospitalier Regional d'Orleans (CHRO) - Hopital La Source, Orléans
  - Hôpital Universitaire Pitié-Salpêtrière, Paris
  - Hopital Europeen Georges-Pompidou, Paris
  - APHP - Hopital Bichat - Claude Bernard, Paris
  - Groupe Hospitalier Diaconesses Croix Saint Simon, Paris
  - Clinical La Croix Du Sud - Ramsay Santé, Quint-Fonsegrives
  - Chu Rennes Hopital Pontchaillou, Rennes
  - Institut de Cancerologie Strasbourg Europe ICANS, Strasbourg
  - CHU Rangueil, Toulouse
- Germany (15):
  - Urologische Partnerschaft Koln UPK, Cologne
  - Urologicum Duisburg, Duisburg
  - Universitatsklinikum Erlangen, Erlangen
  - Universitatsklinikum Essen, Essen
  - Universitaetsklinikum Frankfurt, Frankfurt am Main
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Matthias Schulze - Germany, Markkleeberg
  - Urologie Neandertal Praxis Mettmann, Mettmann
  - Klinikum rechts der Isar an der Technischen Universitat Munchen, München
  - Universitatsklinikum Munster, Münster
  - Klinikum Nurnberg Nord, Nuremberg
  - Medizinisches Versorgungszentrum - Urologie, Nuremberg
  - Studienpraxis Urologie Nurtingen, Nürtingen
  - Caritas-Krankenhaus St. Josef, Regensburg
  - Universitat Tubingen, Tübingen
- India (6):
  - Health Care Global Enterprises pvt Ltd, Bangalore
  - Post Graduate Institute of Medical Education And Research PGIMER, Chandigarh
  - Artemis Hospital, Gurugram
  - Netaji Subhas chandra Bose Cancer Research Institute, Kolkata
  - Tata Memorial Hospital, Mumbai
  - CIMET s Inamdar Multispeciality Hospital, Pune
- Italy (9):
  - Generale Regionale F. Miulli, Acquaviva delle Fonti
  - Ospedale Cardinal Massaia, Asti
  - Ospedale San Giuseppe Moscati di Avellino, Avellino
  - Ospedale San Giacomo Apostolo, Guardia pediatrica territoriale, Castelfranco Veneto
  - Ospedale San Raffaele di Milano, Milan
  - Istituto Europeo di Oncologia, Milan
  - Fondazione G Pascale Istituto Nazionale Tumori IRCCS, Napoli
  - Ospedale S. Maria Delle Croci, Ravenna
  - Istituto Nazionale Tumori Regina Elena, Rome
- Japan (14):
  - Fuji City General Hospital, Fuji-shi
  - Kanazawa University Hospital, Kanazawa
  - Nara Medical University Hospital, Kashihara-shi
  - Kimitsu Chuo Hospital, Kisarazu-shi
  - Kobe City Medical Center General Hospital, Kobe
  - National Hospital Organization Kumamoto Medical Center, Kumamoto
  - Nagano Municipal Hospital, Nagano
  - Nagasaki University Hospital, Nagasaki
  - JRC Nagasaki Genbaku Hospital, Nagasaki
  - Saiseikai Narashino Hospital, Narashino-shi
  - Ehime University Hospital, Toon-shi
  - Toyama University Hospital, Toyama
  - Yamaguchi University Hospital, Ube
  - Yokohama City University Medical Center, Yokohama
- Mexico (5):
  - Consultorio Medico dentro del Hospital Angeles Acoxpa, Mexico City
  - Eme Red Hospitalaria, Mérida
  - Hospital Universitario Dr Jose Eleuterio Gonzalez, Monterrey
  - Avix Investigacion Clinica S C, Monterrey
  - Oncologico Potosino, San Luis Potosí City
- Netherlands (3):
  - Spaarne Ziekenhuis, Hoofddorp
  - Canisius-Wilhelmina Ziekenhuis, Nijmegen
  - Radboud Umcn, Nijmegen
- Poland (9):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - IN VIVO Sp. z o.o, Bydgoszcz
  - Wojewodzki Szpital Specjalistyczny im Stefana Kardynala Wyszynskiego SPZOZ, Lublin
  - Centrum Medyczne, Piotrkow Trybunalski
  - Clinical Research Center sp z o o MEDIC R s k, Poznan
  - Wojewodzki Szpital Specjalistyczny im Janusza Korczaka, Słupsk
  - Provita Poliklinika, Warsaw
  - Narodowy Instytut Onkologii im Marii Sklodowskiej Curie Panstwowy Instytut Badawczy, Warsaw
  - Uniwersytecki Szpital Kliniczny im Jana Mikulicza Radeckiego we Wroclawiu, Wroclaw
- Portugal (3):
  - Ipo Coimbra, Coimbra
  - Uls Santa Maria - Hosp. Santa Maria, Lisbon
  - Uls Gaia Espinho, Vila Nova de Gaia
- South Korea (12):
  - Pusan National University Hospital, Busan
  - Chungbuk National University Hospital, Cheongju-si
  - Kyungpook National University Chilgok Hospital, Daegu
  - Keimyung University Dongsan Hospital, Daegu
  - National Cancer Center, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
- Spain (13):
  - Hosp Univ A Coruna, A Coruña
  - Hosp. Punta de Europa, Algeciras
  - Fund. Puigvert, Barcelona
  - Hosp. Puerta Del Mar, Cadiz
  - Hosp. Gral. Univ. de Castellon, Castellon
  - Hosp. Univ. de Bellvitge, L'Hospitalet de Llobregat
  - Hosp. Univ. Lucus Augusti, Lugo
  - Clinica Univ. de Navarra, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. La Paz, Madrid
  - Hosp Virgen de La Victoria, Málaga
  - Hosp. Univ. Marques de Valdecilla, Santander
  - Hosp. Clinico Univ. de Valencia, Valencia
- Taiwan (6):
  - Kaohsiung Medical University Chung Ho Memorial Hospital, Kaohsiung City
  - Chang Kung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District
- United Kingdom (9):
  - Western General Hospital, Edinburgh
  - St Bartholomews Hospital, London
  - The Royal Marsden NHS Trust, London
  - Charing Cross Hospital, London
  - Derriford Hospital, Plymouth
  - Scunthorpe General Hospital, Scunthorpe
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - Lister Hospital, Stevenage
  - Royal Cornwall Hospitals NHS Trust - Royal Cornwall Hospital, Truro

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency